CLINICAL TRIAL: NCT05955508
Title: Phase 2 Study of Linvoseltamab in Patients With Smoldering Multiple Myeloma at High Risk of Progression to Multiple Myeloma
Brief Title: A Proof-of-Concept Trial to Study the Safety and Activity of Linvoseltamab in Participants With Smoldering Multiple Myeloma at High Risk of Developing Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-2256; 2023-503524-11-00 (Other: EUCT Number)
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Smoldering Multiple Myeloma (SMM)
Keywords: Linvoseltamab; Multiple Myeloma (MM); B cell maturation antigen (BCMA); Bispecific antibody
MeSH Terms: conditions — Smoldering Multiple Myeloma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Safety Run-In (Part 1) (Experimental): Evaluation of initial safety and tolerability of the step-up regimen leading up to the start of full dose linvoseltamab.
  Interventions: Drug: Linvoseltamab
- Expansion (Part 2) (Experimental): Linvoseltamab monotherapy according to the same dosing schedule established in the safety run-in part.
  Interventions: Drug: Linvoseltamab

INTERVENTIONS:
Drug: Linvoseltamab — Administration by intravenous (IV) infusion
  Other Names: REGN5458; Lynozyfic™

SUMMARY:
This study is researching an investigational drug called linvoseltamab ("study drug") in participants at high risk of developing multiple myeloma (MM), a group commonly labeled as high-risk smoldering multiple myeloma (HR-SMM).

The aim of the study is to understand the safety and tolerability (how your body reacts to linvoseltamab) as well as the effectiveness (how well linvoseltamab eliminates plasma cells and prevents the development of MM) of the study drug. There are 2 parts to the study.

* In Part 1, linvoseltamab will be given to a small number of participants to study the early side effects (safety) of the study drug and make sure the treatment is acceptable.
* In Part 2, linvoseltamab will be given to more participants to continue to assess the side effects of the study drug and to evaluate the ability of linvoseltamab to treat HR-SMM and prevent progression to MM.

The study is looking at several other research questions, including:

* How many participants treated with linvoseltamab (study drug) have improvement of their HR-SMM?
* What side effects may happen from taking the study drug?
* How much study drug is in your blood at different times?
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
KEY Inclusion Criteria:

1. High-risk SMM diagnosis within 5 years of study enrollment
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
3. Adequate hematologic and hepatic function, as described in the protocol
4. Estimated glomerular filtration rate ≥30 mL/min/1.73 m^2

KEY Exclusion Criteria:

1. Evidence of myeloma defining events *SLiM CRAB, as described in the protocol

   *SLiM (greater than or equal to Sixty percent clonal plasma cells in the bone marrow, involved/uninvolved free Light chain ratio of ≥100 with the involved free light chain (FLC) being ≥100 mg/L, MRI with >1 focal lesion) CRAB (hyperCalcemia, Renal insufficiency, Anemia, or lytic Bone lesions)
2. Diagnosis of systemic light chain amyloidosis, Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), soft tissue plasmacytoma, or symptomatic multiple myeloma
3. Clinically significant cardiac or vascular disease within 3 months of study enrollment, as described in the protocol
4. Any infection requiring hospitalization or treatment with IV anti-infectives within 28 days of first dose of study drug
5. Uncontrolled human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection; or other uncontrolled infection or unexplained signs of infection
6. History of severe allergic reaction attributed to compounds with a similar chemical or biologic composition as the study drug or excipient

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2032-12-19 (Estimated); Study Completion 2032-12-19 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events of special interest (AESI) during the safety run-in observation period | Up to 35 days
  AESI include grade 2 or higher cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS)
Frequency of treatment-emergent adverse events (TEAEs) during the safety run-in observation period | Up to 35 days
Severity of TEAEs during the safety run-in observation period | Up to 35 days
Complete response (CR) as determined by the investigator | Up to 7 years
Minimal residual disease (MRD) negativity | At 12 months
MRD negativity | At 24 months

SECONDARY OUTCOMES:
Frequency of TEAEs during expansion part | Up to 7 years
  As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Severity of TEAEs during expansion part | Up to 7 years
  As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Frequency of serious adverse events (SAEs) | Up to 7 years
Severity of SAEs | Up to 7 years
Frequency of laboratory abnormalities | Up to 7 years
Severity of laboratory abnormalities | Up to 7 years
Overall response of partial response (PR) or better | Up to 7 years
Duration of response (DOR) | Up to 7 years
Biochemical progression-free-survival (PFS) | Up to 7 years
MRD negativity among participants that achieve very good partial response (VGPR) or better | Up to 3 years after end of treatment
Sustained MRD negativity | Up to 3 years after end of treatment
Time from treatment initiation to date of any myeloma-defining event | Up to 7 years
Time from start of treatment to date of progression to MM or death | Up to 7 years
Time to initiation of first-line treatment for MM | Up to 7 years
Overall survival (OS) | Up to 7 years
Concentration of linvoseltamab in serum over time | Up to 2 years
Incidence of anti-drug antibodies (ADAs) to linvoseltamab over time | Up to 2 years
Titer of ADAs to linvoseltamab over time | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (17):
- Spain (17):
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitari Son Llatzer, Palma Mallorca, Balearic Islands
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar, Murcia
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - University Hospital of Cabuenes, Gijón, Principality of Asturias
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital General Universitario Gregorio Maranon (HGUGM) - Instituto de Investigacion Sanitaria Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - University Hospital Doctor Peset, Valencia
  - La Fe University Hospital, Valencia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/